CLINICAL TRIAL: NCT04955327
Title: A Double-blind, Randomized, Placebo-Controlled, Comparative Study for Assessing the Efficacy and Tolerability of A. Paniculata/A. Chilensis in Individuals With Upper Respiratory Tract Infections
Brief Title: To Compare the Efficacy and Tolerability of A. Paniculata/A. Chilensis in Individuals With URTI
Acronym: A Paniculata
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP/200802/PARACTIN/CC
Record Dates: First submitted 2021-05-05; First posted 2021-07-08 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Andrographis paniculata extract; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A. Paniculata150 mg (Experimental): Extract from Andrographis Paniculata
  Interventions: Drug: A. Paniculata
- A. Chilensis 300 mg (Experimental): Extract from A. Chilensis
  Interventions: Drug: A. Chilensis
- A. Panicluata 150 mg + A. Chilensis 300 mg. (Experimental): combination of extract of A. Paniculata and A. Chilensis
  Interventions: Drug: A. Paniculata and A. Chilensis
- Microcrystalline Cellulose +/-450 mg (Placebo Comparator): Comparator
  Interventions: Drug: Microcrystalline cellulose

INTERVENTIONS:
Drug: A. Paniculata — Extract from A. Paniculata
  Arms: A. Paniculata150 mg
Drug: A. Chilensis — Extract from A. Chilensis
  Arms: A. Chilensis 300 mg
Drug: A. Paniculata and A. Chilensis — Combination of A. Paniculata and A. Chilensis
  Arms: A. Panicluata 150 mg + A. Chilensis 300 mg.
Drug: Microcrystalline cellulose — Placebo comparator
  Arms: Microcrystalline Cellulose +/-450 mg

SUMMARY:
Conventional therapy of upper respiratory tract infection (URTI) is not always effective and sometimes leads to side effects and also to inappropriate use of antibiotic. Hence, a search for safe and effective further treatment options is justified and would be a welcome addition to available conventional treatment. Use of plant based dietary supplements has become increasingly popular over the last few decades or so. Research based on some plants is more than centuries old and its main therapeutic objective is to stimulate the self-healing power of the body. Andrographolide was docked successfully in the binding site of SARS-CoV-2 Mpro. Computational approaches also predicts this molecule to have good solubility, pharmacodynamics property and target accuracy. This molecule also obeys Lipinski's rule, which makes it a promising compound to pursue further biochemical and cell based assays to explore its potential for use against COVID-19. A. Paniculata is a patented extract, standardized to Andrographolide, 14-deoxyandrographolide, and Neo-andrographolide. Maqui contains Maqui Berry Extract of Aristotelia Chilensis (10% Anthocyanidin, 8% Delphinidin) belonging to the family of Elaeocarpaceae, which has been known for its use in several conditions such as sore throat, fever and several other ailments. In the present study, the therapeutic potential of Andrographis Paniculata and Aristotelia chilensis as single ingredients as well as in combination will be evaluated in participants with common cold and COVID related symptoms. The products to be evaluated have been rigorously standardized and are available under the brand names of A. Paniculata and A. Chilensis. Literature indicates that both A. Paniculata and A.Chilensis are effective and safe in the treatment of typical cold-related symptoms in adults.

DETAILED DESCRIPTION:
The common cold is one of the most frequent minor illnesses in the world. A large US-American survey showed that over 70% of the population annually was suffering from at least one viral respiratory tract infection. Also the economic burden in the USA was almost USD 40 billion annually causing considerable direct and indirect healthcare costs. Caused by 200 identified types of viruses, the common cold is primarily associated with rhinoviruses. Common cold symptoms may include sore throat, runny nose, general malaise, and low-grade fever at onset, followed by nasal congestion and cough. While benign, they last for several days and cause 40% of all missed work days. Complications also include sinusitis, otitis media and pneumonia, exacerbations of asthma and chronic obstructive pulmonary disease, and serious illness in immunocompromised patients.

Colds typically afflict most adults and adolescents 2-4 times a year and symptoms usually peak around day 3 or 4 and last 1-2 weeks with a median of 7 days. There is no approved specific therapy for URTI, treatment is therefore mainly symptomatic. The most common pharmacological treatments are antipyretics, anti-inflammatory drugs, expectorants, decongestants, and cough suppressants, either alone or in combination. Supportive measures can include bed rest, hot baths, and inhalations, gargling, and drinking plenty of fluids. Antibiotics are widely prescribed, but often is inappropriate because URTI are mostly caused by viruses and are only indicated in the case of bacterial infection. Its overuse can also lead to the development of community acquired resistant pathogens which are an increasing and serious health burden.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged between 18 and 50 years, complete as of the screening date.
2. Participants with symptoms of acute upper respiratory tract infection as assessed by the investigator at the time of screening.
3. Participants with BMI ≤ 29.9 kg/m2.
4. Upper respiratory tract infection symptoms present for at least 24 hours but not more than 72 hours prior to screening visit.
5. Those having a score of ≥ 5 for at least 2 symptoms out of runny nose, plugged nose, sneezing, sore throat, scratchy throat, cough or head congestion on the Wisconsin Upper Respiratory Symptom Survey-21.
6. Participants not requiring hospitalization.
7. Participants with COVID +ve/ COVID -ve RT-PCR report.
8. SPO2 level ≥ 90%
9. Systolic blood pressure < 130 mm Hg and/or diastolic blood pressure < 90.
10. Those who demonstrate an understanding of the study details and have a willingness to participate, as evidenced by voluntary written informed consent.
11. Must be literate and have the ability to complete the study-based questionnaires and requirements.

Exclusion Criteria:

1. High grade fever defined as body temperature ≥ 40°C.
2. With a history of allergy (allergic rhinitis) along with symptoms such as sneezing, runny nose and red, watery and itchy eyes.
3. Chest X-ray showing signs of pneumonia.
4. Participants with history of chronic obstructive pulmonary disease, pulmonary fibrosis or asthma
5. Participants with rhinitis medicamentosa, chronic cough of bacterial, fungal or other known origin.
6. Participants with anatomical nasal obstruction/ deformity or nasal reconstructive surgery etc.
7. Participants with history of heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies.
8. Participants with history of immunocompromised state immune system with/ without organ transplant.
9. Participants with known or suspected hypersensitivity or intolerance to herbal products.
10. Alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 2.0 times the upper limit of normal.
11. Participants diagnosed with Sickle cell disease, Thalassemia, Type I/ II diabetes mellitus, cystic fibrosis.
12. Diagnosed cases of hypertension.
13. Those not willing to abstain from home based cold remedies that include but are not limited to steam inhalation, decoctions, vapour rub, ginger tea, honey tea, decoctions, or any form of dietary supplements during the entirety of study participation period.
14. Those who have been vaccinated for influenza, swine flu or COVID three months prior to screening visit.
15. Those who have taken or should be taking or are taking antibiotics, antivirals, steroids, nasal decongestants, antihistamines or other medications that are expected to alleviate cold symptoms within one week of the start of the study.
16. Those who have severe mental illnesses, such as dementia, Parkinson's disease, Alzheimer's Disease, depression or anxiety disorders, or those who are currently taking psychoneurological drugs, such as antidepressants.
17. Those who have participated in other clinical trials within 30 days, prior to the screening visit or plan to participate in other clinical trials during the trial period.
18. Participants with substance abuse as per last two year history that includes the use of but is not limited to drugs such as cocaine, amphetamine, marijuana etc.
19. Individuals having a history of smoking or currently smoking or using any form of smokeless tobacco.
20. Participants with heavy alcohol consumption, defined as:

    1. For men: More than 14 standard alcoholic drink (SAD)/week or more than 4 SAD in a day.
    2. For women: More than 7 SAD/week or more than 3 SAD in a day.
    3. Binge drinkers, defined as 5 or more SAD for men, in a 2-hour time frame.
    4. Binge drinkers, defined as 4 or more SAD for Women, in a 2-hour time frame. (NOTE - A standard alcoholic drink contains approximately 14 grams of alcohol, which is equivalent to 12 ounces of beer (~5% alcohol), 8.5 ounces of malt liquor (~9% alcohol), 5 ounces of wine (~12% alcohol), 3.5 ounces of fortified wine (e.g., sherry or port), or 1.5 ounces of liquor (distilled spirits; ~40% alcohol)
21. Those who have clinically significant disorder/s of cardiovascular, endocrine, lymphatic, respiratory, hepatobiliary, urinary, reproductive, central nervous system, musculoskeletal and digestive systems.
22. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
23. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Severity Outcome | Day 0, 1, 2, 3, 4, 5, 6, and 7
  Change in total symptom severity scores from 0 to 7 (where 0 means not sick to 7 means severe) as assessed by Wisconsin Upper Respiratory Symptom Survey-21 on day 7 from baseline and in comparison to placebo.

SECONDARY OUTCOMES:
Time to resolve symptoms | Day 0, 1, 2, 3, 4, 5, 6, and 7
  Time to resolution of common cold like symptoms as assessed by participant reporting '0 = not sick' out of 7, for any one day during treatment period as per Wisconsin Upper Respiratory Symptom Survey-21
percentage wise severity resolution | 7 days
  Percentage of participants with resolved common cold like complaints at the end of day 7 in comparison to placebo (unresolved participants being those who do not report "0 = not sick" out of 7, as per Wisconsin Upper Respiratory Symptom Survey-21, till the end of treatment period.
Minimal Important Difference | Day 0, 5, and 7
  Percentage of participants achieving minimal important difference of ≥ 10.3 Wisconsin Upper Respiratory Symptom Survey-21 total scores at day 5 and 7 from baseline and in comparison to placebo. Therefore, in the study Minimal important difference will be calculated as the difference of Wisconsin Upper Respiratory Symptom Survey-21 total scores from baseline to day 5 and day 7 and if it is ≥ 10.3, it will be deemed as clinically significant treatment effect.
Visual Analogue Scale based severity outcomes | Day 0, 1, 2, 3, 4, 5, 6, and 7
  Change in participant's fever and burning eyes sensation severity scores (from 0 to 7 where 0 means not at all severe to 100 means very severe) as assessed by visual analogue scale on day 7 from baseline and in comparison to placebo.
Change in symptom resolution | Day 0 to day 7 (for all COVID +ve participants) and Day 8 to day 15 (For COVID participants who didn't turn negative on day 8)
  Change in severity of COVID related symptoms (from 0 to 7 where 0 means no symptom to 7 means severe) as assessed by total scores of COVID diary at day 7 and day 15 from baseline and in comparison to placebo.

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - St . George Hospital, Mumbai, Maharashtra
  - Gillurkar Multispecialty Hospital, Nagpur, Maharashtra
  - Shree Hospital & Critical Care Center, Nagpur, Maharashtra
  - Apollo Spectra Hospitals, Kanpur, Uttar Pradesh
  - Shubham Sudbhawana Super Specialty Hospital, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No